CLINICAL TRIAL: NCT03149627
Title: Chronic Hepatitis B Virus Clinical Epidemiology in a Representative Sample of Zambian Adults
Acronym: HEP-ZED
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital (Unknown); Tropical Gastroenterology and Nutrition Group (Unknown); Centre for Infectious Disease Research in Zambia (Other); Ministry of Health, Zambia (Other Government)
Responsible Party: Principal Investigator, Michael Vinikoor, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: X160524001
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2019-01

CONDITIONS: HBV; Alcoholic Hepatitis; Liver Fibroses
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Part 1: The Investigators will test for active HBV infection using a rapid point-of-care HBsAg test. In addition, as a service to clients who have not had an HIV test in the past year (as recommended by Ministry of Health), for 10% of participants (selected randomly at household level), the Investigators will also collect a dried blood spot using finger prick method to perform HBcAb test, an epidemiologic test for lifetime exposure to HBV.
  Part 2: Participants will have physical examination, a liver ultrasound, transient elastography (TE), and blood will be collected for HBV viral load and other markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals from selected households: Individuals residing in selected households in Lusaka Province, Zambia.
  Interventions: Other: Estimates - prevalence of lifetime/chronic HBV infection

INTERVENTIONS:
Other: Estimates - prevalence of lifetime/chronic HBV infection — Estimation of the prevalence and correlates of lifetime HBV infection defined as hepatitis B core antibody (HBcAb) positivity and chronic HBV infection defined as HBsAg positivity.

SUMMARY:
The purpose of this study is to recruit a random and representative sample of individuals within several Zambian communities for markers of Hepatitis B Virus (HBV) and to characterize chronic HBV infection and indications for treatment.

DETAILED DESCRIPTION:
The Zambian Ministry of Health (MoH) considers viral hepatitis a significant public health threat; however, there are limited representative data on HBV burden, risk factors, clinical significance, and interaction with co-infections and co-morbidities that are common in Zambia. In collaboration with the Central Statistical Office, MoH, and Centers for Disease Control and Prevention, the Zambia Population-Based HIV Impact Assessment (ZAMPHIA) will be testing a representative sample of Zambians across all 10 provinces for HBV infection. This is an important first step toward understanding the burden of disease and its distribution across the country. The goal of this study is to generate further information for consumption by local and regional health policymakers. The Investigators will research the epidemiologic risk factors for lifetime and current HBV infection, characterize clinical features of chronic HIV in Zambia, and describe key virological, serological, and comorbid factors that are critical to developing the best policies for HBV control in Zambia.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: 18 years or older, current residence in selected household
* Part 2: Participant in part 1 of the study, HBsAg-positive by rapid point-of-care test

Exclusion Criteria:

* Part 1: Unable to provide informed consent
* Part 2: Unwilling to travel to a hospital in their province

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1: 6,000 individuals residing in randomly selected households in Lusaka Province in Zambia regardless of the clinically health status.
  Part 2: All part 1 participants who test HBsAg-positive (anticipated sample size of 250) during community testing.
Sampling Method: Non-Probability Sample
Enrollment: 5003 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Prevalence and correlates of lifetime HBV infection | baseline
  Estimates of the prevalence and correlates of lifetime HBV infection defined as hepatitis B core antibody (HBcAb) positivity and chronic HBV infection defined as HBsAg positivity in randomly selected households in Lusaka Province in Zambia. Identification of individual (such as age or sex) and community (such as province) correlates of lifetime and chronic HBV infection.

SECONDARY OUTCOMES:
Proportion of Zambian adults who require antiviral therapy for chronic HBV infection | within 1 month of part 1
  Estimate the proportion of Zambian adults who require antiviral therapy for chronic HBV infection in randomly selected households in Lusaka Province in Zambia.
Clinical phenotypes of patients with chronic HBV infection | within 1 month of part 1
  Determining clinical phenotypes (such as chronic active or inactive) of patients with chronic HBV infection.
Frequency of primary drug resistance mutations. | within 1 month of part 1
  Frequency of primary drug resistance mutations.
The proportion of patients with chronic HBV infection who have significant liver fibrosis or cirrhosis. | within 1 month of part 1
  Estimate the proportion of patients with chronic HBV infection who have significant liver fibrosis or cirrhosis using non-invasive tests.
Unhealthy alcohol use in HBV-positive patients | within 1 month of part 1
  Proportion of unhealthy alcohol users measured with the Alcohol Use Disorders Identification Test, and the association of unhealthy alcohol use with liver fibrosis markers among patients with chronic HBV infection. Among participants in part 2 of the study, the Investigators will also describe the prevalence of unhealthy drinking using data from the AUDIT-C screen. The Investigators will categorize patients as 'unhealthy drinkers' if the AUDIT-C score is >3 for men and >2 for women. The Investigators will also assess hepatosplenic schistosomiasis, defined by grade 2 or grade 3 periportal liver fibrosis on abdominal ultrasound. The Investigators will use bivariable and multivariable regression to compare liver fibrosis markers by AUDIT-C score (non/moderate drinkers versus unhealthy drinkers).
Hepatosplenic schistosomiasis co-infection with liver fibrosis markers among patients with chronic HBV infection | within 1 month of part 1
  Hepatosplenic schistosomiasis co-infection with liver fibrosis markers among patients with chronic HBV infection. The Investigators will also assess hepatosplenic schistosomiasis, defined by grade 2 or grade 3 periportal liver fibrosis on abdominal ultrasound. The Investigators will use bivariable and multivariable regression to compare liver fibrosis markers by the presence of hepatosplenic schistosomiasis.
HIV prevalence in HBV-patients | within 1 month of part 1
  HIV prevalence in HBV-patients by self-report or rapid test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Vinikoor, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided